CLINICAL TRIAL: NCT04252235
Title: A Randomized Controlled Trial of Home Air Purification for Eosinophilic COPD
Brief Title: Home Air Purification for Eosinophilic COPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Mary Rice, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P001129
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: COPD; Eosinophilia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Eosinophilia | interventions — Air Filters

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive real or sham HEPA filters in the bedroom and living room for a total of 12 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sham air purifiers will be indistinguishable from real air purifiers. Only the research assistant installing the purifiers and the data coordinating center will have knowledge of assignment to real or sham purifiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham air purifier (Sham Comparator): Participants will receive a sham air purifier that will be installed in the bedroom and living room. These purifiers will make a noise, but will not filter the air.
  Interventions: Device: Sham air purifier
- True air purifier (Experimental): Participants will receive a HEPA air purifier in the bedroom and living room.
  Interventions: Device: Air purifier

INTERVENTIONS:
Device: Air purifier — The intervention is the placement of active HEPA air purifiers in the bedroom and living room of the true air purifier arm. These air purifiers have been shown to reduce levels of particles in the home.
  Arms: True air purifier
Device: Sham air purifier — The intervention is the placement of sham HEPA air purifiers in the bedroom and living room. These purifiers look identical to real HEPA air purifiers, but do not filter the air.
  Arms: Sham air purifier

SUMMARY:
This study evaluates the influence of home air purification on the lung health of adults with eosinophilic COPD. Half of the participants will receive real air purifiers (HEPA filters) and half will receive sham air purifiers.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the third most common cause of death in the United States, and is exacerbated by exposure to air pollution. Knowledge about whether air purification affects the health of those with eosinophilic COPD (approximately 40% of all COPD patients seeking care), who generally have more active airway inflammation. If found to be beneficial, home air purification may offer a non-pharmacologic intervention for a large proportion of people with this common and serious disease.

This study will evaluate whether home air purification affects lung function, respiratory symptoms, nasal biomarkers (inflammatory proteins and metals) among people with eosinophilic COPD. Participants will be randomized to receive real or sham air purifier in the bedroom and living room for 12 months. The intervention group will receive two high efficiency particulate air (HEPA) air purifiers, while the control group will receive two sham air purifiers that look and sound the same as real HEPA air purifiers.

ELIGIBILITY:
Inclusion Criteria:

* Age of 40 years or more
* Physician diagnosis of COPD [Global Initiative for Obstructive Lung Disease (GOLD) Stage II-IV disease with Forced Expiratory Volume (FEV1)/ Forced Vital Capacity (FVC) ≤70% and FEV1 (% predicted) <80%]
* Blood eosinophil count of >=150 cells per μL at screening or in the previous year
* Former smoker with tobacco exposure of >=10 pack-years

Exclusion Criteria:

* Inability to complete monthly questionnaires
* Inability to perform lung function testing
* Regularly using a portable HEPA air purifier in the home at time of enrollment
* End stage chronic disease with life expectancy <2 years as determined by PI judgment
* Living in location other than home (e.g. long term care facility)
* Planning to change residence within the study period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in forced expiratory volume in 1 second (FEV1) | Baseline [3 months before intervention and day of intervention] and post intervention [7 days, 6 months and 12 months]
  FEV1 is the volume of air exhaled in the first second of a forced exhalation maneuver. Lower volumes indicate worse lung function.

SECONDARY OUTCOMES:
Change in health status (also called health-related quality of life) by St. George Respiratory Questionnaire | Baseline [3 months before intervention and day of intervention] and post-intervention [6 months and 12 months]
  The St. George's Respiratory Questionnaire is scored from 0 to 100. Higher scores indicate more health impairment.
Change in respiratory symptoms | Monthly for 3 months preintervention and 12 months post-intervention
  The Breathlessness, Cough and Sputum Scale measures the severity of respiratory symptoms in COPD. The total score ranges from 0 to 12, with higher scores indicating greater symptom severity.
Change in functional capacity by 6 minute walk test | The 6 minute walk test measures distance (in meters) walked in a time of 6 minutes
  Baseline and 12 months post-intervention

OTHER OUTCOMES:
Change in nasal inflammatory mediators | Baseline [3 months before intervention and day of intervention] and post intervention [7 days, 6 months and 12 months]
  Concentrations of inflammatory mediators relevant to allergic and non-allergic airway pathophysiology will be measured repeatedly at baseline and post-randomization in the nasal lining fluid by nasosorption. Mediators will include including Eotaxin, Eotaxin-3, GM-CSF, IFN-γ, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IL-10, IL-12/IL-23p40, IL-12p70, IL-13, IL-15, IL-16, IL-17A, IP-10, MCP-1, MCP-4, MDC, MIP-1α, MIP-1β, TARC, TNF-α, TNF-β, VEGF-A

CONTACTS AND LOCATIONS:
Overall Officials: Mary B Rice, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
After study completion, data requests for post-hoc analyses may be submitted to the PI who will discuss each request with members of the research team and External Advisory Committee. If approved, we will facilitate secure access to data with appropriate coding files that will allow interpretation of the dataset. We will utilize data-sharing agreements to restrict the transfer of data, requiring that data be used only for research purposes. If excessive data preparation is needed, we will request funds from the requester to cover the additional personnel and resource costs.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After study completion, requests for data sharing will be addressed within 3 months.
Access Criteria: Data requests must be accompanied by a data analysis plan, which includes the scientific background and rationale for the proposed analysis, variables needed, analytical approach, and qualifications of the research team. Investigators must be able to demonstrate they have the skills and resources to analyze the data and protect the data in a secure environment.

REFERENCES:
- [Derived] Saeed MS, Denoncourt CM, Chao IA, Schortmann S, Nassikas NJ, Synn AJ, Koutrakis P, Coull BA, Kang CM, Wolfson JM, Ferguson ST, Rebuli ME, Jaspers I, Liu JP, Greco KF, Phipatanakul W, Rice MB. Protocol for the air purification for eosinophilic COPD study (APECS): a randomised controlled trial of home air filtration by HEPA. BMJ Open. 2024 Jan 18;14(1):e074655. doi: 10.1136/bmjopen-2023-074655. PMID 38238060